CLINICAL TRIAL: NCT04683588
Title: Effect of Continuous Nursing Care Applied to Total Knee Arthroplasty Patients With Coaching Strategy on Some Patient Outcomes: Randomized Controlled Trial
Brief Title: The Effect of Coaching Strategy on Some Patient Outcomes After Total Knee Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Melike Durmaz, Nurse, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 93804542-020
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Pain; Anxiety; Self Efficacy; Patient Satisfaction; Lifestyle-related Condition
Keywords: Nursing coaching; Postoperative care; Total Knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Patient Satisfaction; Mental Disorders

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized controlled study to determine the pre- and postoperative nursing care patients' anxiety level, pain control, self-care capacity, nursing care service and hospital re-hospitalization in patients who underwent total knee prosthesis
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): 1. Polyclinic: Pre-tests (pain, anxiety, self-care and daily living activities), General coaching, 60 minutes
  2. Before Surgery: Nursing coaching, 30-45 minutes
  3. Surgery Day: Nursing coaching, 30-45 minutes
  4. Postoperative 1st Day: Nursing coaching, 30-45 minutes
  5. Postoperative 2nd Day: Nursing coaching practice, 30-45 minutes
  6. Day of discharge: Nursing coaching, 30-45 minutes.
  7. 15 days after discharge: Nursing coaching, 60 minutes
  8. 45 days after the operation: Nursing coaching, 60 minutes.
  9. 90 days after surgery: Nursing coaching, 60 minutes.
  Interventions: Other: Nursing Coaching
- Control arm (No Intervention): Patients in the control group will receive routine postoperative nursing care.

INTERVENTIONS:
Other: Nursing Coaching — Different strategies, methods and training techniques are used in the implementation of preoperative and postoperative nursing care of surgical patients scheduled for total knee arthroplasty surgery. One of them is patient coaching. Coaching is a method that increases the quality of nursing care.While the coaching strategy contributes more to the recovery process of the patient with the role of the case manager of the nurse, it provides a reduction in the problems related to surgery (pain, nausea-vomiting, mobilization problems), reduction in repeated hospitalizations and positive contributions to the cost.
  Arms: intervention arm

SUMMARY:
Total knee arthroplasty (TKA); It is frequently applied to adults, especially those over the age of 55. Total knee arthroplasty surgery is among the surgeries with a high satisfaction rate for the patient, although complications can develop and this rate varies between 1.65-11.3%. It has a privileged place in the prevention, early diagnosis and treatment of the problems and complications that may occur. In this way, patients' anxiety will be reduced, self-care competence will be provided, recovery process will be accelerated, quality of life and care satisfaction will increase. In this context, the training, information, skill-building, counseling and care practice that the nurse will provide to the patient; With the results to be obtained from this study, patients with TKA can be given pre-operative and post-operative nursing care using a nurse coaching strategy, and patients' anxiety level, pain control, patient satisfaction It is predicted to have a positive effect on self-care ability and re-hospitalization rates. Thus, it is thought that both quality healthcare services will be provided and will contribute to the creation of evidence-based data. It is thought that the study will also contribute to the dissemination of the pre-operative and postoperative nurse coaching strategy in patients undergoing TKA, and will guide the planning of nursing education. This study is an experimental study to determine the effect of continuous nursing care given with a coaching strategy to patients scheduled for TKA surgery on anxiety, pain, self-care ability, satisfaction, and re-hospitalization. The study will be carried out in Konya Private Hospital. Data collection time is set as September-December 2020. Data will be collected by the researcher using the Diagnostic questionnaire form, State Anxiety Scale, Visual Analog Scale, Newcastle Nursing Care Satisfaction Scale, Modified Barthel index and Self-Care Ability Scale. In this context, the training, information, skill-building, counseling and care practice that the nurse will provide to the patient; It will contribute to achieving the desired results by positively affecting both the success of the surgery and the healing process of the patient.

DETAILED DESCRIPTION:
The universe of the research; patients who are planned to undergo total knee arthroplasty between January 1, 2021 and June 1, 2021 in the orthopedic surgery clinic where the study will be conducted will comprise the patients who meet the inclusion criteria and agree to participate in the study. The research was planned as a randomized controlled experimental study. Block randomization method will be used to determine the experimental and control groups. In order for the groups to be distributed homogeneously, the order produced by a computer program (www.randomizer.org) will be used. Randomization will be done by a biostatistician outside the researcher. Patients who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental and control groups according to the randomization list. Research data will be collected in a hospital's orthopedics and traumatology service surgery ward between 1 January 2021 - 1 June 2021.

The dependent variables of the study are postoperative statue anxiety score, patient self-care ability score, pain severity (Visual Analog Scale-VAS), pain control and status ( pain-causing conditions, analgesic such as use case), patient satisfaction score, re-hospitalization average. In the research, "Individual Characteristics Form" and "Patient Follow-up Form" prepared by the researcher in line with the literature will be used as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

Being literate, Turkish speaking and verbal communication, Absence of cognitive diseases such as Alzheimer's, delirium and dementia, No psychiatric problems, Being 18 years or older, Living in Konya city center

Exclusion Criteria:

Having undergone a revision total knee replacement operation, Application of analgesic medication to the knee joint space during surgery, Application of patient controlled analgesia (PCA) in postoperative pain control, Not understanding the content of the research, Having a health problem that prevents exercising or evaluating,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Postoperative pain severity | Reported pain severity in the first 24 hours after surgery
  Pain severity assessment with Visual Assessment Scale (VAS) Score: 0-10; 0- No Pain, 10- Worst pain
Postoperative self-care ability scale | Reported self-care ability status in the first 24 hours after surgery
  Self -care ability scale with score: 0-5; 0-lowest, 5-highest
state anxiety scale | Reported self-care ability status in the first 24 hours after surgery
  state anxiety scale score :1-4 ; 1-Lowest , 4-Highest
New Castle Nursing Care Satisfaction | Postoperative will be evaluated 72. hour.
  New Castle Nursing Care Satisfaction Scale:1-5 1-Lowest , 5-Highest
Modified Barthel index | After the outpatient clinic examination evaluation(preoperative); 72. hour after surgery; 15th day after discharge; 45 days after discharge; 90th day after discharge.
  Modified Barthel index 0-15 0-Lowest, 15 Highest

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Kurşun, PhD, Principal Investigator — ŞEYH ŞAMİL NEIGHBORHOOD DOSTELİ AVENUE NO: 52/1 SELÇUKLU / KONYA (BEHİND SELÇUKLU MUNİCİPALİTY)
Locations (1):
- Medova Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No